CLINICAL TRIAL: NCT07307846
Title: Investigation of the Effects of Interlaminar Epidural Steroid Injection on Upper Extremity Proprioception in Patients With Chronic Cervical Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Marmara-FTR-GNY-03
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cervical Radiculopathy; Cervical Radicular Pain; Proprioception
Keywords: cervical radiculopathy; cervical radicular pain; interlaminar epidural steroid injection; proprioception; proprioceptive impairment
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cervical Radiculopathy- Interlaminar Epidural Steroid Injection (ILESI) Group (Active Comparator): Participants diagnosed with chronic unilateral cervical radiculopathy due to cervical disc herniation will undergo a standardized interlaminar epidural steroid injection. All evaluations (proprioception, pain, neuropathic pain, disability, grip strength, and quality of life) will be performed at baseline (T0), 3 weeks post-procedure (T1), and 3 months post-procedure (T2).
  Interventions: Procedure: Interlaminar Epidural Steroid Injection (ILESI)

INTERVENTIONS:
Procedure: Interlaminar Epidural Steroid Injection (ILESI) — The injection will be administered under sterile conditions with fluoroscopic guidance at the C7-T1 interlaminar level. An 18-gauge epidural needle will be advanced into the epidural space, followed by injection of a mixture containing: 80 mg triamcinolone acetonide, 1 mL of 2% lidocaine, and 2 mL of 0.9% saline.
  Participants will remain under observation for approximately 2 hours after the procedure and will then be discharged. The procedure will be performed by an experienced pain medicine specialist with over 15 years of fluoroscopic interventional practice.

SUMMARY:
Cervical radiculopathy is a common condition caused by irritation or compression of cervical nerve roots, often leading to unilateral neuropathic pain and functional impairment. Proprioceptive deficits in the upper extremity have been demonstrated in various cervical spine disorders; however, the effect of interlaminar epidural steroid injection (ILESI) on upper extremity proprioception in patients with chronic cervical radiculopathy has not been previously examined.

This prospective interventional study aims to evaluate changes in upper extremity proprioception following unilateral ILESI in patients with cervical disc herniation-related chronic radiculopathy. A secondary aim is to investigate the relationship between proprioceptive changes and clinical outcomes such as pain, neuropathic pain, disability, grip strength, and quality of life.

DETAILED DESCRIPTION:
Cervical radiculopathy is characterized by neuropathic pain radiating along a dermatomal pattern due to irritation or compression of cervical nerve roots, most commonly from cervical disc herniation or foraminal narrowing. In addition to sensory symptoms, proprioceptive deficits may arise from altered cervical afferent input, affecting upper extremity joint position sense and sensorimotor control. Although proprioceptive impairment has been previously demonstrated in chronic neck pain and cervical spondylosis, the proprioceptive profile of patients with cervical radiculopathy has not been adequately investigated.

Interlaminar epidural steroid injection (ILESI) is a commonly used minimally invasive treatment for cervical disc herniation-associated radicular pain and has been shown to reduce pain and improve function and disability. However, its potential effects on upper extremity proprioception, an important sensory component contributing to coordinated movement and rehabilitation outcomes, remain unknown.

This prospective interventional study will evaluate proprioceptive changes using the PRO-Reach upper extremity joint position sense test, a validated multi-planar assessment method that measures joint position error across multiple directions without requiring computerized or robotic devices. Clinical outcome measures will include neuropathic pain scores, pain intensity, disability indices, hand-grip strength, and health-related quality of life. All assessments will be performed at three time points: before treatment (T0), 3 weeks after injection (T1), and 3 months after injection (T2).

Participants will undergo standardized unilateral ILESI at the C7-T1 interlaminar level under fluoroscopic guidance using a combination of corticosteroid, local anesthetic, and saline. Data collection will be performed by blinded assessors to minimize measurement bias.

The study aims to characterize whether ILESI provides measurable improvements in upper extremity proprioception and to determine the extent to which changes in proprioceptive accuracy correspond to changes in pain, neuropathic symptoms, upper extremity function, and quality of life. These findings may help guide rehabilitation planning and provide insight into the sensorimotor consequences of cervical radiculopathy and its interventional treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following:

* Female or male, 18-65 years of age
* Presence of unilateral cervical radicular pain lasting at least 3 months
* MRI of the cervical spine within the last 12 months demonstrating at least one cervical disc herniation consistent with the patient's symptoms
* Diagnosed with chronic cervical radiculopathy based on history, physical examination, and clinical evaluation
* Ability to read and write (literacy)
* Willingness to participate and ability to provide written informed consent

Exclusion Criteria:

Participants will be excluded for any of the following:

* Cervical physical therapy or cervical spinal injection performed within the past 6 months
* Symptoms or diagnosis of upper extremity entrapment neuropathy
* Documented vitamin B12 deficiency or vitamin D deficiency on laboratory results within the past year
* History of cervical spine surgery or significant cervical trauma
* Bilateral cervical radicular pain
* Cervical spinal stenosis
* History of upper extremity surgery or significant upper extremity trauma
* Cognitive impairment, major psychiatric disorder, intellectual disability, or history of significant neurological disease
* Diagnosis of polyneuropathy
* Diagnosis of Diabetes Mellitus
* Diagnosis of fibromyalgia
* Current use of medications that may impair proprioception or have sedative effects (e.g., gabapentinoids, antidepressants, muscle relaxants)
* Active local or systemic infection
* Coagulopathy or bleeding diathesis
* Known allergy to any components of the planned injection (triamcinolone, lidocaine, saline, contrast medium)
* Pregnancy
* Inability or unwillingness to provide informed consent
* Illiteracy (unable to read or write)

Withdrawal Criteria

* Voluntary withdrawal of consent at any time
* Inability or unwillingness to continue study participation for any reason
* New medical condition or event after enrollment that renders continuation unsafe according to the investigator's judgment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Upper Extremity Proprioception Error (PRO-Reach) | Baseline (T0), 3 weeks after ILESI (T1), and 3 months after ILESI (T2)
  Upper extremity joint position sense will be assessed using the PRO-Reach test, which quantifies position error (distance in centimeters between the target and reproduced position) across multiple reaching directions. The primary outcome is the change in mean position error of the affected upper extremity between baseline and follow-up assessments. Higher values indicate poorer proprioceptive accuracy.

SECONDARY OUTCOMES:
Change in Neuropathic Pain Score (DN-4) | Baseline (T0), 3 weeks after ILESI (T1), and 3 months after ILESI (T2)
  Neuropathic pain symptoms will be evaluated using the Douleur Neuropathique 4 (DN-4) questionnaire. Scores range from 0 to 10, with scores ≥4 indicating the presence of neuropathic pain. The outcome is the change in DN-4 score over time.
Change in Pain Intensity (Numeric Rating Scale, NRS 0-10) | Baseline (T0), 3 weeks after ILESI (T1), and 3 months after ILESI (T2)
  Pain intensity related to cervical radicular pain will be measured using an 11-point Numeric Rating Scale (NRS), where 0 represents "no pain" and 10 represents "worst imaginable pain." Neck and extremity pain will be recorded as two separate subscores. The outcome is the change in NRS score over time. Lower scores indicate less pain.
Change in Health-Related Quality of Life (SF-12) | Baseline (T0), 3 weeks after ILESI (T1), and 3 months after ILESI (T2)
  Health-related quality of life will be assessed using the 12-Item Short Form Survey (SF-12), generating physical and mental component summary scores. Higher scores indicate better perceived health status, ranging between 0-100. The outcome is the change in SF-12 scores over time.
Change in Hand-Grip Strength (kg) | Baseline (T0), 3 weeks after ILESI (T1), and 3 months after ILESI (T2)
  Maximal isometric hand-grip strength will be measured using a dynamometer (e.g., Jamar) with the participant seated, elbow at 90° flexion, and wrist in neutral. Three trials will be performed for each hand, and the mean value will be recorded in kilograms. The outcome is the change in grip strength of the affected side over time. Higher values indicate greater strength.
Change in Upper Extremity Function (QuickDASH Score) | Baseline (T0), 3 weeks after ILESI (T1), and 3 months after ILESI (T2)
  Upper extremity function and disability will be evaluated using the Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire. Scores range from 0 to 100, with higher scores indicating greater disability. The outcome is the change in QuickDASH score over time.

CONTACTS AND LOCATIONS:
Overall Officials: Savaş Şencan, Assoc. Prof., Pain Medicine, Study Director — Algology Division, Department of Physical Medicine and Rehabilitation, Marmara University Faculty of Medicine
Locations (1):
- Marmara University Pendik Training and Research Hospital, Pendik, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documents will be available 6 months after publication of the main results and remain accessible for at least 5 years following publication.
Access Criteria: Qualified researchers may request access to the de-identified dataset and supporting documentation by submitting a brief research proposal and data access agreement to the corresponding investigator (Gökçenur Yalçın, M.D., Department of Physical Medicine and Rehabilitation, Marmara University, Istanbul, Turkey). Data will be shared via a secure institutional data repository upon approval by the principal investigator and the Marmara University Ethics Committee.